CLINICAL TRIAL: NCT03557775
Title: Respiratory Muscle Strength Training in Presbyphonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00064753
Record Dates: First submitted 2018-05-22; First posted 2018-06-15 (Actual); Results first posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-08

CONDITIONS: Presbylarynx
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Perceptual ratings of voice quality and of videostroboscopic images of the larynx will be rater by external judges, who will be blinded to the group assignment and to the assessment time (pre or post treatment).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Inspiratory Muscle Strength Training (Experimental): The participants in the IMST arm will receive, in addition to standard of care voice therapy, inspiratory muscle strength training (IMST).
  The IMST intervention will consist of 5 sets of 5 breaths in the inspiratory threshold device every day during four weeks, with a loading dose set at 75% of the participants' maximal inspiratory pressure (MIP). MIP will be measured once a week during the weekly supervised session to adjust the inspiratory trainer.
  Interventions: Device: Inspiratory Muscle Strength Training (IMST); Behavioral: Voice Exercises
- Expiratory Muscle Strength Training (Experimental): The participants in the EMST arm will receive, in addition to standard of care voice therapy, expiratory muscle strength training (EMST).
  The EMST intervention will consist of 5 sets of 5 breaths in the expiratory threshold device every day during four weeks, with a loading dose set at 75% of the participants' maximal expiratory pressure (MEP). MEP will be measured once a week during the weekly supervised session to adjust the inspiratory trainer.
  Interventions: Device: Expiratory Muscle Strength Training (EMST); Behavioral: Voice Exercises
- Voice Exercises (Active Comparator): The participants in the voice exercises group will receive standard of care voice therapy with a speech language pathologist, once a week during four weeks, plus daily practices.
  Interventions: Behavioral: Voice Exercises

INTERVENTIONS:
Device: Inspiratory Muscle Strength Training (IMST) — IMST will be conducted using an inspiratory pressure threshold trainer (Philips Respironics® Threshold IMT or POWERbreathe® Medic Plus), which consists of a mouthpiece with a spring-loaded valve. The valve blocks the airflow until the threshold pressure is achieved by breathing in forcefully into the device. This allows airflow as long as the sufficient pressure is maintained.
  Other Names: Inspiratory muscle training (IMT); Respiratory muscle training (RMT); Respiratory muscle strength training (RMST); Philips Respironics® Threshold IMT; POWERbreathe® Medic Plus
  Arms: Inspiratory Muscle Strength Training
Device: Expiratory Muscle Strength Training (EMST) — EMST will be conducted using an expiratory pressure threshold trainer (EMST150®), which consists of a mouthpiece with a spring-loaded valve. The valve blocks the airflow until the threshold pressure is achieved by breathing out forcefully into the device. This allows airflow as long as the sufficient pressure is maintained.
  Other Names: Expiratory muscle training (EMT); Respiratory muscle training (RMT); Respiratory muscle strength training (RMST); EMST150®
  Arms: Expiratory Muscle Strength Training
Behavioral: Voice Exercises — Voice exercises will consist of the Vocal Function Exercises (VFE) protocol, developed by Stemple (2005). It contains 4 steps: (a) sustain the vowel /i/ on the musical note F for as long as possible. Repeat as judged by the SLP. (b) Glide from the lowest note to the highest note. Repeat as judged by the SLP. (c) Glide from the highest note to the lowest note. Repeat as judged by the SLP. (d) Sustain the notes C-D-E-F-G for as long as possible. Each note will be repeated until the participant finds the right placement (forward-focused voice), as judged by the SLP. Humming will be used to facilitate placement.

SUMMARY:
Presbyphonia is an age-related voice disorder that affects more than 10 million people in the United States. Presbyphonia is characterized by vocal fold atrophy that impairs older individuals' ability to communicate, leading to social isolation and reduced quality of life. Outcomes from current treatment approaches are often suboptimal for patients with presbyphonia as they do not sufficiently challenge the respiratory system to induce meaningful change. It is highly likely that the addition of respiratory training would result in greatly improved outcomes, such as the ability to speak loud and long enough to have a normal conversation. The purpose of this study will be to examine the effect of adding inspiratory muscle strength training (IMST) or expiratory muscle strength training (EMST) to standard of care voice therapy on respiratory and voice outcomes in patients with an age-related voice disorder.

Forty-eight participants diagnosed with presbyphonia will be blocked-randomized into three intervention groups, using a 3-parallel arm design: IMST and voice exercises, EMST and voice exercises, and voice exercises during all session. Study endpoints will be the change in voice and respiratory measures after four treatment sessions compared to baseline values. Response to treatment will be analyzed to determine if there are subgroups of high- or low-responders based on baseline voice and respiratory characteristics.

ELIGIBILITY:
Inclusion Criteria:

* must receive a diagnosis of presbyphonia by a trained laryngologist. The diagnosis will be given following a visual examination if the observations are consistent with the characteristics of a presbylarynx, as judged by the laryngologist.
* must be 50 years old and older.

Exclusion Criteria:

* has received voice therapy in the past year
* presents with a vocal fold pathology other than presbyphonia
* has a known neurologic or a progressive neuromuscular disease
* has a medical condition that could be aggravated by the experimental intervention, or any condition judged by the physician (Dr. Halstead) as being unsuitable for RMST.
* has dysarthria or a language disorder
* has a hearing loss that is not adequately managed
* has a cognitive disorder that might affect treatment compliance
* is unable to give informed consent

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Bonilha, PhD, Principal Investigator — Medical University of South Carolina; Maude Desjardins, M.Sc., Study Director — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: We had 22 subjects enrolled, however one did not meet the screening requirements and was not further included in the study (and therefore was not randomized to an intervention group). Another participant withdrew before being randomized to an intervention group. In total, 20 participants were randomized to the intervention groups.
Groups:
- Inspiratory Muscle Strength Training: The participants in the IMST arm will receive, in addition to standard of care voice therapy, inspiratory muscle strength training (IMST).
- Expiratory Muscle Strength Training: The participants in the EMST arm will receive, in addition to standard of care voice therapy, expiratory muscle strength training (EMST).
Period: Overall Study
Arm/Group | Inspiratory Muscle Strength Training | Expiratory Muscle Strength Training | Voice Exercises
Started | 5 | 7 | 8
Completed | 4 | 4 | 4
Not Completed | 1 | 3 | 4
Not completed — Withdrawal by Subject | 1 | 2 | 4
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Considering the pilot data of the study, the study team enrolled even participants who would not be able to complete the study protocol because of transportation burden. However, the study team considered only participants who COMMITTED to the whole protocol for baseline and results analysis. Only data for those subjects are presented here.
Groups:
- Total: Total of all reporting groups
Arm/Group | Inspiratory Muscle Strength Training | Expiratory Muscle Strength Training | Voice Exercises | Total
Number analyzed (Participants) | 4 | 4 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.50 (8.74) | 70.50 (7.23) | 77.50 (4.66) | 71.83 (7.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 1 | 5
  Male | 1 | 3 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 4 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 4 | 4 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 4 | 12
Reflux Symptom Index score [Mean (Standard Deviation); unit: Score on a scale] — The Reflux Symptom Index score can range from 0 to 45, with a lower score considered a more favorable outcome. A score greater than 13 is associated with a reflux-related issue.
  Score on a scale | 19.75 (3.59) | 14.50 (5.80) | 14.25 (8.54) | 16.17 (6.29)
Voice Handicap Index score [Mean (Standard Deviation); unit: Score on a scale] — The Voice Handicap Index score can range from 0 to 40, with a lower score being more favorable. A score greater than 11 is indicative of a voice-related handicap.
  Score on a scale | 24.00 (6.06) | 13.75 (7.93) | 21.25 (6.19) | 19.67 (7.62)

OUTCOME MEASURES:

1. Primary Outcome: Post-Treatment Mean in Voice Handicap Index Score
Description: Voice Handicap Index-10 (ordinal scale that measures the degree of handicap a person experiences because of their voice disorder. Minimum score 0, maximal score 40. A lower score is better )
Time Frame: up to 5 weeks after baseline
Population: Per protocol
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inspiratory Muscle Strength Training | Expiratory Muscle Strength Training | Voice Exercises
Number analyzed (Participants) | 4 | 4 | 4
score on a scale | 15.00 (4.97) | 15.75 (8.77) | 18.50 (10.66)
Statistical Analysis 1: Comparison: Inspiratory Muscle Strength Training vs Expiratory Muscle Strength Training vs Voice Exercises; Null hypothesis: there will be no significant time by group interaction effect for this variable; Test type: Superiority; p = 0.041, ANOVA — Result for time by group interaction (threshold for statistical significance set at 0.05)

2. Secondary Outcome: Post-treatment Mean in (Habitual) Sound Pressure Level
Description: Acoustic measure of loudness, in Decibels
Time Frame: up to 5 weeks after baseline
Population: Per protocol
Measure: Mean (Standard Deviation); unit: Decibels (dB)
Arm/Group | Inspiratory Muscle Strength Training | Expiratory Muscle Strength Training | Voice Exercises
Number analyzed (Participants) | 4 | 4 | 4
Decibels (dB) | 73.18 (5.29) | 70.73 (1.65) | 74.75 (2.60)
Statistical Analysis 1: Comparison: Inspiratory Muscle Strength Training vs Expiratory Muscle Strength Training vs Voice Exercises; Null hypothesis: there will be no significant time by group interaction effect for this variable; Test type: Superiority; p = 0.887, ANOVA — Result for time by group interaction. Statistical threshold set at 0.05

3. Secondary Outcome: Post-treatment Mean in Baseline Smoothed Cepstral Peak Prominence (CPPS) (During Reading)
Description: Acoustic measure of voice quality, in Decibels
Time Frame: up to 5 weeks after baseline
Population: Per protocol
Measure: Mean (Standard Deviation); unit: Decibels (dB)
Arm/Group | Inspiratory Muscle Strength Training | Expiratory Muscle Strength Training | Voice Exercises
Number analyzed (Participants) | 4 | 4 | 4
Decibels (dB) | 18.03 (1.83) | 16.74 (0.52) | 17.86 (1.06)
Statistical Analysis 1: Comparison: Inspiratory Muscle Strength Training vs Expiratory Muscle Strength Training vs Voice Exercises; Null hypothesis: there will be no significant time by group interaction effect for this variable; Test type: Superiority; p = 0.733, ANOVA — Result for time by group interaction effect. Threshold for statistical significance was set at 0.05

4. Secondary Outcome: Post-treatment Mean in Baseline Noise-to-harmonic Ratio (NHR)
Description: Acoustic measure of voice quality, expressed as a ratio of noise to harmonics in the signal.
Time Frame: up to 5 weeks after baseline
Population: Per protocol
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Inspiratory Muscle Strength Training | Expiratory Muscle Strength Training | Voice Exercises
Number analyzed (Participants) | 4 | 4 | 4
ratio | 0.13 (0.02) | 0.16 (0.06) | 0.12 (0.01)
Statistical Analysis 1: Comparison: Inspiratory Muscle Strength Training vs Expiratory Muscle Strength Training vs Voice Exercises; Null hypothesis: there will be no significant time by group interaction effect for this variable; Test type: Superiority; p = 0.702, ANOVA — Result for time by group interaction effect. Threshold for statistical significance set at 0.05

5. Secondary Outcome: Post-Treatment Mean in Baseline Amplitude Perturbation Quotient (APQ)
Description: Acoustic measure of voice quality, expressed as a percentage
Time Frame: up to 5 weeks after baseline
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Inspiratory Muscle Strength Training | Expiratory Muscle Strength Training | Voice Exercises
Number analyzed (Participants) | 4 | 4 | 4
percentage | 2.91 (1.04) | 4.25 (2.56) | 3.05 (0.60)
Statistical Analysis 1: Comparison: Inspiratory Muscle Strength Training vs Expiratory Muscle Strength Training vs Voice Exercises; Null hypothesis: there will be no significant time by group interaction effect for this variable; Test type: Superiority; p = 0.198, ANOVA — Result for time by group interaction effect. Threshold for statistical significance set at 0.05

6. Secondary Outcome: Post-treatment Mean in Overall Severity of Voice Quality
Description: This is a auditory-perceptual measure rated on the standardized form: Consensus Auditory-Perceptual Evaluation of Voice (a 100-mm visual analogue scale where 0 represents a normal voice and 100 represents an extremely disrupted voice quality. A lower score is better).
Time Frame: up to 5 weeks after baseline
Population: Per protocol
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Inspiratory Muscle Strength Training | Expiratory Muscle Strength Training | Voice Exercises
Number analyzed (Participants) | 4 | 4 | 4
units on a scale | 21.00 (10.61) | 31.25 (28.65) | 35.00 (17.78)
Statistical Analysis 1: Comparison: Inspiratory Muscle Strength Training vs Expiratory Muscle Strength Training vs Voice Exercises; Null hypothesis: there will be no significant time by group interaction effect for this variable; Test type: Superiority; p = 0.388, ANOVA — Result for time by group interaction effect. Threshold for statistical significance set at 0.05

7. Secondary Outcome: Post-treatment Mean in Baseline Bowing Index
Description: Measure of vocal fold atrophy, calculated as the length of the membranous vocal fold/distance from the edge x100. The index was calculated based on still images from the larynx obtained from videostroboscopy. A smaller bowing index is indicative of less atrophy, and is therefore a better outcome. A greater bowing index is indicative of more atrophy and represent a worse outcome.
Time Frame: up to 5 weeks after baseline
Population: Per protocol
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Inspiratory Muscle Strength Training | Expiratory Muscle Strength Training | Voice Exercises
Number analyzed (Participants) | 4 | 4 | 4
Index | 9.03 (3.35) | 5.76 (0.96) | 8.97 (1.05)
Statistical Analysis 1: Comparison: Inspiratory Muscle Strength Training vs Expiratory Muscle Strength Training vs Voice Exercises; Null hypothesis: there will be no significant time by group interaction effect for this variable; Test type: Superiority; p = 0.296, ANOVA — Result for time by group interaction effect. Threshold for statistical significance set at 0.05

8. Secondary Outcome: Post-treatment Mean in Communicative Participation Item Bank (CPIB) Score
Description: Ordinal scale measuring the impact of the communication disorder on various situations. A higher score is indicative of a more functional communication (the minimum score is 0 and the maximum score is 30).
Time Frame: up to 5 weeks after baseline
Population: Per protocol
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inspiratory Muscle Strength Training | Expiratory Muscle Strength Training | Voice Exercises
Number analyzed (Participants) | 4 | 4 | 4
score on a scale | 24.00 (1.00) | 19.50 (7.14) | 14.75 (7.27)
Statistical Analysis 1: Comparison: Inspiratory Muscle Strength Training vs Expiratory Muscle Strength Training vs Voice Exercises; Null hypothesis: there will be no significant time by group interaction effect for this variable; Test type: Superiority; p = 0.040, ANOVA — Result for time by group interaction effect. Threshold for statistical significance set at 0.05

9. Secondary Outcome: Post-treatment Mean in Glottal Function Index (GFI) Score
Description: Glottal Function Index (ordinal scale that measures the presence and degree of symptoms of glottal dysfunction experienced by a patient. Minimum score is 0, maximum score is 20. A lower score is better).
Time Frame: up to 5 weeks after baseline
Population: Per protocol
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Inspiratory Muscle Strength Training | Expiratory Muscle Strength Training | Voice Exercises
Number analyzed (Participants) | 4 | 4 | 4
score on a scale | 9.75 (4.03) | 8.75 (4.27) | 8.75 (5.50)
Statistical Analysis 1: Comparison: Inspiratory Muscle Strength Training vs Expiratory Muscle Strength Training vs Voice Exercises; Null hypothesis: there will be no significant time by group interaction effect for this variable; Test type: Superiority; p = 0.887, ANOVA — Result for time by group interaction effect. Threshold for statistical significance set at 0.05

10. Secondary Outcome: Post-treatment Mean in Average Glottal Airflow
Description: Aerodynamic measure of voice expressed in Liters/second
Time Frame: up to 5 weeks after baseline
Population: Per protocol
Measure: Mean (Standard Deviation); unit: liters/second
Arm/Group | Inspiratory Muscle Strength Training | Expiratory Muscle Strength Training | Voice Exercises
Number analyzed (Participants) | 4 | 4 | 4
liters/second | 0.10 (0.06) | 0.27 (0.06) | 0.18 (0.08)
Statistical Analysis 1: Comparison: Inspiratory Muscle Strength Training vs Expiratory Muscle Strength Training vs Voice Exercises; Null hypothesis: there will be no significant time by group interaction effect for this variable; Test type: Superiority; p = 0.663, ANOVA — Result for time by group interaction effect. Threshold for statistical significance was set 0.05

11. Secondary Outcome: Post-treatment Mean in Average Subglottal Pressure
Description: Aerodynamic measure of voice expressed in cmH20
Time Frame: up to 5 weeks after baseline
Population: Per protocol
Measure: Mean (Standard Deviation); unit: cmH20
Arm/Group | Inspiratory Muscle Strength Training | Expiratory Muscle Strength Training | Voice Exercises
Number analyzed (Participants) | 4 | 4 | 4
cmH20 | 6.37 (2.33) | 6.47 (1.96) | 5.99 (0.32)
Statistical Analysis 1: Comparison: Inspiratory Muscle Strength Training vs Expiratory Muscle Strength Training vs Voice Exercises; Null hypothesis: there will be no significant time by group interaction effect for this variable; Test type: Superiority; p = 0.026, ANOVA — Result for time by group interaction effect. Threshold for statistical significance set at 0.05

12. Secondary Outcome: Post-treatment Mean in Aerodynamic Resistance
Description: Aerodynamic measure (subglottal pressure divided by mean flow rate), expressed as cmH20/liters/second
Time Frame: up to 5 weeks after baseline
Population: Per protocol
Measure: Mean (Standard Deviation); unit: cmH20/liters/second
Arm/Group | Inspiratory Muscle Strength Training | Expiratory Muscle Strength Training | Voice Exercises
Number analyzed (Participants) | 4 | 4 | 4
cmH20/liters/second | 63.43 (17.07) | 21.25 (7.71) | 37.11 (15.11)
Statistical Analysis 1: Comparison: Inspiratory Muscle Strength Training vs Expiratory Muscle Strength Training vs Voice Exercises; Null hypothesis: there will be no significant time by group interaction effect for this variable; Test type: Superiority; p = 0.721, ANOVA — Result for time by group interaction effect. Threshold for statistical significance set at 0.05

13. Secondary Outcome: Post-treatment Mean in Maximum Expiratory Pressure (MEP)
Description: Indirect measure of respiratory (expiratory) muscle strength, expressed in cmH20
Time Frame: up to 5 weeks after baseline
Population: Per protocol
Measure: Mean (Standard Deviation); unit: cmH20
Arm/Group | Inspiratory Muscle Strength Training | Expiratory Muscle Strength Training | Voice Exercises
Number analyzed (Participants) | 4 | 4 | 4
cmH20 | 121.00 (69.29) | 176.25 (25.85) | 131.00 (40.60)
Statistical Analysis 1: Comparison: Inspiratory Muscle Strength Training vs Expiratory Muscle Strength Training vs Voice Exercises; Null hypothesis: there will be no significant time by group interaction effect for this variable; Test type: Superiority; p = 0.408, ANOVA — Result for time by group interaction effect. Threshold for statistical significance set at 0.05

14. Secondary Outcome: Post-treatment Mean in Maximum Inspiratory Pressure (MIP)
Description: Indirect measure of respiratory muscle strength, expressed in cmH20
Time Frame: up to 5 weeks after baseline
Population: Per protocol
Measure: Mean (Standard Deviation); unit: cmH20
Arm/Group | Inspiratory Muscle Strength Training | Expiratory Muscle Strength Training | Voice Exercises
Number analyzed (Participants) | 4 | 4 | 4
cmH20 | 98.75 (43.49) | 84.50 (18.91) | 81.50 (9.82)
Statistical Analysis 1: Comparison: Inspiratory Muscle Strength Training vs Expiratory Muscle Strength Training vs Voice Exercises; Null hypothesis: there will be no significant time by group interaction effect for this variable; Test type: Superiority; p = 0.638, ANOVA — Result for time by group interaction effect. Threshold for statistical significance set at 0.05

15. Secondary Outcome: Post-treatment Mean in Forced Vital Capacity (FVC)
Description: Measure of pulmonary function, expressed as a percent predicted value
Time Frame: up to 5 weeks after baseline
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percentage of predicted value
Arm/Group | Inspiratory Muscle Strength Training | Expiratory Muscle Strength Training | Voice Exercises
Number analyzed (Participants) | 4 | 4 | 4
percentage of predicted value | 80.75 (20.87) | 80.75 (22.81) | 94.00 (10.46)
Statistical Analysis 1: Comparison: Inspiratory Muscle Strength Training vs Expiratory Muscle Strength Training vs Voice Exercises; Null hypothesis: there will be no significant time by group interaction effect for this variable; Test type: Superiority; p = 0.715, ANOVA — Result for time by group interaction effect. Threshold for statistical significance set at 0.05

16. Secondary Outcome: Post-treatment Mean in Forced Expiratory Volume in 1 Second (FEV1)
Description: Measure of pulmonary function expressed as percent predicted value
Time Frame: up to 5 weeks after baseline
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percentage of predicted value
Arm/Group | Inspiratory Muscle Strength Training | Expiratory Muscle Strength Training | Voice Exercises
Number analyzed (Participants) | 4 | 4 | 4
percentage of predicted value | 75.75 (20.76) | 73.00 (32.44) | 94.00 (8.91)
Statistical Analysis 1: Comparison: Inspiratory Muscle Strength Training vs Expiratory Muscle Strength Training vs Voice Exercises; Null hypothesis: there will be no significant time by group interaction effect for this variable; Test type: Superiority; p = 0.708, ANOVA — Result for time by group interaction effect. Threshold for statistical significance set at 0.05

17. Secondary Outcome: Post-Treatment Mean for FEV1/FVC
Description: Pulmonary function measure expressed as percent predicted value (ratio between forced expiratory volume in one second and forced vital capacity)
Time Frame: up to 5 weeks after baseline
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percentage of predicted value
Arm/Group | Inspiratory Muscle Strength Training | Expiratory Muscle Strength Training | Voice Exercises
Number analyzed (Participants) | 4 | 4 | 4
percentage of predicted value | 94.00 (4.69) | 87.75 (20.12) | 99.00 (2.94)
Statistical Analysis 1: Comparison: Inspiratory Muscle Strength Training vs Expiratory Muscle Strength Training vs Voice Exercises; Null hypothesis: there will be no significant time by group interaction effect for this variable; Test type: Superiority; p = 0.988, ANOVA — Result for time by group interaction effect. Threshold for statistical significance set at 0.05

18. Other Pre Specified Outcome: Voice-Vibratory Assessment With Laryngeal Imaging
Description: exploratory measure
Time Frame: up to 5 weeks after baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Inspiratory Muscle Strength Training | Expiratory Muscle Strength Training | Voice Exercises
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/7 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 1/5 | 1/7 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Inspiratory Muscle Strength Training (N=5) | Expiratory Muscle Strength Training (N=7) | Voice Exercises (N=8)
Skin irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — The participant reported the presence of marks on the lips that seemed to have been caused by the mouthpiece of the muscle pressure meter, potentially because of a sucking effect during inspiratory muscle strength testing. The marks were temporary.
Transient aching (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — One participant reported transient aching in the ribcage after doing IMST. The participant's aching resolved. The study team lowered the load on the device and the participant was told to stop the exercises if feeling any aching.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-26): https://cdn.clinicaltrials.gov/large-docs/75/NCT03557775/Prot_SAP_000.pdf